CLINICAL TRIAL: NCT01733485
Title: Electrophilic Fatty Acid Derivatives in Asthma
Acronym: EFADA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sally E. Wenzel MD (Other)
Responsible Party: Sponsor-Investigator, Sally E. Wenzel MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: U10HL098177 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Asthma; Electrophilic Fatty Acids
Keywords: Asthma; Electrophilic Fatty Acids; Inflammation
MeSH Terms: conditions — Asthma; Inflammation | interventions — Aspirin; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aspirin (Active Comparator)
  Interventions: Drug: Aspirin
- Indomethacin (Active Comparator)
  Interventions: Drug: Indomethacin
- Control (No Intervention)

INTERVENTIONS:
Drug: Aspirin — 500 mg/8 h for 5 days
  Arms: Aspirin
Drug: Indomethacin — 25 mg/8 h for 5 days
  Arms: Indomethacin

SUMMARY:
Asthma is an inflammatory disease, which means it causes swelling in the lungs to cause shortness of breath and/or wheezing. There are several asthma medications that help to reduce this problem.

The objective of this research study is to characterize the presence of electrophilic fatty acids in the bronchial airway of subjects with controlled asthma at baseline and after treatment with Aspirin, Indomethacin, or no treatment at all. The presence of electrophilic fatty acids may indicate inflammation. Aspirin and Indomethacin are known to respectively increase and inhibit the formation of electrophilic fatty acids. By gaining a better understanding of how electrophilic fatty acids work and how they respond to different treatment, researchers hope to be able to find better ways to lessen airway inflammation in asthma in the future.

DETAILED DESCRIPTION:
Relevant to asthma, the chemical identities and potent anti-inflammatory signaling actions of endogenously-produced Electrophilic Fatty acid OXidation products (EFOXs) have recently been described. Endogenous EFOXs include nitro and alpha and beta-unsaturated ketone derivatives of unsaturated fatty acids that are generated as byproducts of a) fatty acid oxidation and nitration by inflammatory-derived reactive species and b) enzymatic fatty acid oxygenation reactions catalyzed by cyclooxygenase-2 and lipoxygenases. Recent data reveal that multiple salutary post-translational protein modifications are induced by EFOXs. Specifically, the covalent adduction of functionally-significant thiols in signaling proteins occurs, with these reactions modulating critical inflammatory signaling pathways. These signaling proteins include the nuclear lipid receptor PPARg and the redox-sensitive transcription factors NF kappaB and Keap1/Nrf2. This proposed research investigates the concept that the reversible reaction of EFOXs with critical transcription factors results in the regulation of adaptive responses to inflammation.

In this clinical study, bronchoalveolar lavage fluid (BAL) will be obtained from asthmatics treated with COX-2 inhibitors that enhance (aspirin) and inhibit (indomethacin) COX-2 dependent EFOX generation, as well as from those assigned to no intervention. BAL will be obtained from healthy, non-smoking adults with controlled asthma having at least a 12% increase in FEV1 after short-acting bronchodilator treatment or a positive methacholine response (reduction in FEV1 ≥ 20% at or before 16 mg/ml). A total of 30 asthmatic subjects will be randomized (10 per arm) to a) aspirin, b) indomethacin or c) no intervention groups

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate asthma
* No evidence of a previous asthma exacerbation in the preceding 6 weeks (defined as increased severity of respiratory symptoms requiring systemic steroids or escalation of therapy; b) asthma control questionnaire (ACQ) score less than 1.

Exclusion Criteria:

* Diagnosis of severe asthma, vocal cord dysfunction, cystic fibrosis, COPD, CAD, hypertension, diabetes or renal failure that is not well controlled
* Greater than 10 pack-year history of smoking;
* Stopped smoking less than 1 year prior to study,
* Taking any aspirin or other NSAIDS on the week prior to bronchoscopy,
* Taking omega-3 fatty acid supplements
* If a subject is currently taking an omega-3 fatty acid supplement and is interested in the study, after a 30 day wash out, the participant can be re-screened and evaluated for participation.
* Taking pioglitazone or rosiglitazone (synthetic thiazolidinedione PPARg ligands);
* other known pulmonary diseases;
* Inability to undergo bronchoscopy,
* Contraindications or allergy to aspirin or indomethacin,
* Asthmatics with known hypersensitivity to aspirin, and
* Steroid (systemic) dependent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2016-09 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Airway concentration of electrophilic fatty acids | Change in the bronchoalveolar lavage concentration of electrophilic fatty acids from the first to the second bronchoscopy
  Patients undergo a baseline bronchoscopy, afterwhich they are randomized to 5 days of a)indomethacin, b) aspirin, c) nothing . After treatment, another bronchoscopy is done. Outcomes are determined after each bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States